CLINICAL TRIAL: NCT02756572
Title: A Feasibility Study of "Early" Allogeneic Hematopoietic Cell Transplantation for Relapsed or Refractory High-Grade Myeloid Neoplasms
Brief Title: Early Allogeneic Hematopoietic Cell Transplantation in Treating Patients With Relapsed or Refractory High-Grade Myeloid Neoplasms
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Mary-Beth Percival, Assistant Professor, Division of Hematology, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9567; NCI-2016-00477 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9567 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH); RG1016011 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2016-04-21; First posted 2016-04-29 (Estimated); Results first posted 2021-03-22 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-10

CONDITIONS: Blasts 10 Percent or More of Bone Marrow Nucleated Cells; Chronic Myelomonocytic Leukemia-2; High Grade Malignant Neoplasm; Myelodysplastic Syndrome; Myelodysplastic Syndrome With Excess Blasts-2; Myeloid Neoplasm; Previously Treated Myelodysplastic Syndrome; Recurrent Acute Myeloid Leukemia; Refractory Acute Myeloid Leukemia
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute | interventions — Cladribine; Cyclosporine; Cyclosporins; Cytarabine; Filgrastim; Granulocyte Colony-Stimulating Factor; fludarabine phosphate; Melphalan; Mitoxantrone; Mycophenolic Acid; Sirolimus; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (chemotherapy, HCT) (Experimental): See Detailed Description
  Interventions: Drug: Cladribine; Drug: Cyclosporine; Drug: Cytarabine; Biological: Filgrastim; Drug: Fludarabine Phosphate; Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Other: Laboratory Biomarker Analysis; Drug: Melphalan; Drug: Mitoxantrone Hydrochloride; Drug: Mycophenolate Mofetil; Other: Questionnaire Administration; Drug: Sirolimus; Radiation: Total-Body Irradiation; Drug: Melphalan Hydrochloride

INTERVENTIONS:
Drug: Cladribine — Given IV
  Other Names: 2-CdA; 2CDA; CdA; Cladribina; Leustat; Leustatin; Leustatine; RWJ-26251
Drug: Cyclosporine — Given PO
  Other Names: 27-400; Ciclosporin; CsA; Cyclosporin; Cyclosporin A; Gengraf; Neoral; OL 27-400; Sandimmun; Sandimmune; SangCya
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Biological: Filgrastim — Given SC
  Other Names: FILGRASTIM, LICENSE HOLDER UNSPECIFIED; G-CSF; Neupogen; r-metHuG-CSF; Recombinant Methionyl Human Granulocyte Colony Stimulating Factor; rG-CSF; Tevagrastim
Drug: Fludarabine Phosphate
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; SH T 586
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Undergo allogeneic hematopoietic stem cell transplantation
  Other Names: Allogeneic Hematopoietic Stem Cell HSCT; Allogeneic Stem Cell Transplantation; HSC
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Melphalan — Given IV
  Other Names: Alanine Nitrogen Mustard; CB-3025; L-PAM; L-Phenylalanine Mustard; L-sarcolysin; L-Sarcolysin Phenylalanine mustard; L-Sarcolysine; Melphalanum; Phenylalanine Mustard; Phenylalanine nitrogen mustard; Sarcoclorin; Sarkolysin; WR-19813
Drug: Mitoxantrone Hydrochloride — Given IV
  Other Names: CL 232315; DHAD; DHAQ; Dihydroxyanthracenedione Dihydrochloride; Mitoxantrone Dihydrochloride; Mitoxantroni Hydrochloridum; Mitozantrone Hydrochloride; Mitroxone; Neotalem; Novantrone; Onkotrone; Pralifan
Drug: Mycophenolate Mofetil — Given PO
  Other Names: Cellcept; MMF
Other: Questionnaire Administration — Ancillary studies
Drug: Sirolimus — Given PO
  Other Names: AY 22989; RAPA; Rapamune; Rapamycin; SILA 9268A; WY-090217
Radiation: Total-Body Irradiation — Undergo TBI
  Other Names: Total Body Irradiation; Whole-Body Irradiation
Drug: Melphalan Hydrochloride — Given IV
  Other Names: 241286; 3-(p-(bis(2-chloroethyl)amino)phenyl)-L-Alanine; Hydrochloride; Alkeran; Alkerana; Evomela

SUMMARY:
This clinical trial studies how well early stem cell transplantation works in treating patients with high-grade myeloid neoplasms that has come back after a period of improvement or does not respond to treatment. Drugs used in chemotherapy, such as filgrastim, cladribine, cytarabine and mitoxantrone hydrochloride, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving chemotherapy before a donor peripheral blood cell transplant helps stop the growth of cells in the bone marrow, including normal blood-forming cells (stem cells) and cancer cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. The donated stem cells may also replace the patient's immune cells and help destroy any remaining cancer cells. Early stem cell transplantation may result in more successful treatment for patients with high-grade myeloid neoplasms.

DETAILED DESCRIPTION:
OUTLINE:

RE-INDUCTION CHEMOTHERAPY: Patients receive filgrastim subcutaneously (SC) on days 0-5, mitoxantrone hydrochloride intravenously (IV) over 60 minutes on days 1-3, cladribine IV over 2 hours on days 1-5, and cytarabine IV over 2 hours on days 1-5.

CONDITIONING REGIMEN: Beginning 14-60 days after re-induction chemotherapy, patients receive fludarabine phosphate IV over 30 minutes on days -6 to -2, melphalan IV on days -3 to -2, cyclosporine orally (PO) twice daily (BID) starting on day -3. Sirolimus PO BID starting on day -3 will be given to patients who have matched unrelated donors or mismatched unrelated donors. Patients >55 years or with significant co-morbidities will only receive melphalan IV on day -2 and will also receive total body irradiation (TBI) on day -1 or day 0.

EARLY TRANSPLANT: Patients undergo allogeneic HCT after conditioning regimen on day 0.

GVHD PROPHYLAXIS: Patients with matched donors will receive mycophenolate mofetil PO three times daily (TID) on days 0-30, then twice a day (BID) until day 40; and cyclosporine PO BID on days -3 to 96, with a taper until day 150. Patients with matched unrelated donors also receive sirolimus PO BID on days -3 to 150, with a taper until day 180. Patients with mismatched unrelated donors will receive mycophenolate mofetil PO TID on days 0-30, then BID until day 100, with a taper until day 150; cyclosporine PO BID on days -3 to 150, then taper until day 180; and sirolimus BID PO days -3 to 180, then a taper until day 365.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

INCLUSION CRITERIA (ENROLLMENT)

* Relapsed or refractory high-grade myeloid neoplasms, defined as having a blast count of >= 10% blasts at initial diagnosis; examples include excess blasts (EB)-2, with >= 10% blasts at initial diagnosis, acute myeloid leukemia (AML) or chronic myelomonocytic leukemia (CMML-2); standard definitions of relapse will apply (i.e., characterized by >= 5% abnormal blasts or blast equivalents as assessed by multiparameter flow cytometry or morphologic examination; peripheral blood blasts or blast equivalents; or extramedullary granulocytic sarcoma, per European LeukemiaNet [ELN] 2017 guidelines); bone marrow aspirate/biopsy will be accepted if performed outside University of Washington/Fred Hutchinson Cancer Research Center (UW/FHCRC); determination of disease status should occur within 30 days of signing informed consent

  * R/R high-grade myeloid neoplasm following intensive induction chemotherapy; relapsed high-grade myeloid neoplasm: patients will be classified as relapsed if they have >= 5% blasts after being in a complete remission (CR) following treatment for high-grade myeloid neoplasm; refractory high-grade myeloid neoplasm: patients may be classified as refractory if they have received at least one prior cycle of induction chemotherapy, whether with cladribine cytarabine mitoxantrone (GCLAM) or another regimen

    ** Patients may have received up to two courses of intensive induction chemotherapy during initial treatment prior to enrollment on this protocol; for example, patients who have received two courses of granulocyte colony stimulating factor (G-CSF) GCLAM (or similar) chemotherapy, with most recent high-dose cytarabine-containing chemotherapy > 6 months ago and CR lasting > 6 months, will be eligible for this protocol; regimens "similar to GCLAM" would include cytarabine at doses of 1g/m^2 for at least 5 doses; examples of regimens "similar to GCLAM" would be GCLA, fludarabine cytarabine granulocyte (FLAG), and FLAG-idarubicin (ida); however, patients who received more than two courses of GCLAM (or similar) chemotherapy, or patients who received two courses of GCLAM and had CR lasting < 6 months, would not be eligible
  * R/R high-grade myeloid neoplasm following less intensive induction chemotherapy. Patients who have received at least three cycles of treatment with a hypomethylating agent (HMA; such as azacitidine or decitabine) and still have >= 10% blasts will be eligible for the study (they will be considered refractory); similarly, patients who have received three or more cycles of HMA therapy who have had a response (e.g., achieving CR with < 5% blasts), but who then progress using standard definitions of relapse, will also be eligible (they will be considered relapsed)
* Potentially eligible for reduced intensity conditioning based on known organ function (formal organ function testing may occur after consent)
* Caregiver capable of providing post-HCT care
* Written informed consent

INCLUSION CRITERIA (TRANSPLANT)

* Identified donor (see DONOR SELECTION below for further details)

  * Matched related or unrelated (one allele mismatch in HLA-A, B, or C OK) donor according to institutional standards
  * Unrelated volunteer donor who is mismatched with the recipient (i.e. 9/10 match)
* Caregiver capable of providing post-HCT care, who will be present once induction therapy with filgrastim, cladribine, cytarabine, mitoxantrone hydrochloride (GCLAM) begins
* Written informed consent for transplant
* Either bone marrow or peripheral blood is allowed

Exclusion Criteria:

EXCLUSION CRITERIA (ENROLLMENT)

* Prior allogeneic HCT
* More than two prior courses of induction chemotherapy
* Relapse after minimal residual disease (MRD)-negative CR within 3 months of most recent GCLAM chemotherapy
* Low likelihood of being eligible for reduced intensity conditioning HCT based on known information

  * Cardiac ejection fraction < 40% or symptomatic coronary artery disease or uncontrolled arrhythmia, as assessed by multigated acquisition (MUGA) or transthoracic echocardiography (TTE) within previous 3 months and since the most recent anthracycline exposure
  * Corrected diffusing capacity of the lungs for carbon monoxide (DLCOc) < 40% or forced expiratory volume in 1 second (FEV1) < 50%
  * Estimated glomerular filtration rate (GFR) < 40 ml/min
  * Need for supplemental oxygen
  * Direct bilirubin or alanine aminotransferase (ALT) > 2 x upper limit of normal, unless these abnormalities are thought to be related to Gilbert's disease or leukemic infiltration of hepatic parenchyma
* Known human immunodeficiency virus (HIV) positivity
* Pregnant or nursing (to be confirmed with quantitative human chorionic gonadotropin [HCG] testing)
* Invasive solid tumor within 5 years; non-melanoma skin cancer or in situ malignancies are allowed
* Evidence of serious uncontrolled infection
* Eastern Cooperative Oncology Group (ECOG) of 3 or 4
* EXCLUSION CRITERIA (TRANSPLANT)
* Donor specific antibodies against donor HLA-DQ or -DP
* Active bacterial, fungal or viral infections unresponsive to medical therapy
* Active leukemia in the central nervous system (CNS)
* HIV positive
* Cardiac ejection fraction < 40% or symptomatic coronary artery disease or uncontrolled arrhythmia
* DLCOc < 40% or FEV1 < 50%
* Estimated GFR < 40 ml/min
* Need for supplemental oxygen
* Direct bilirubin or ALT > 2 x upper limit of normal, unless these abnormalities are thought to be related to Gilbert's disease or leukemic infiltration of hepatic parenchyma

DONOR SELECTION:

Identification of an appropriate donor will follow the general guidelines listed below.

* HLA-matched related or unrelated donor. Donors must be:

  * Matched for HLA-A, B, C, DRB1 and DQB1 by high resolution typing
  * Only a single allele disparity will be allowed for HLA-A, B, or C as defined by high resolution typing
* HLA-mismatched unrelated donor. Unrelated volunteer donors who are mismatched with the recipient within one of the following limitations will be permitted:

  * Mismatch for one HLA class I antigen with or without an additional mismatch for one HLA-class I allele, but matched for HLA-DRB1 and HLA-DQ, OR
  * Mismatched for two HLA class I alleles, but matched for HLA-DRB1 and HLA-DQ
  * HLA class I HLA-A, -B, -C allele matched donors allowing for any one or two DRB1 and/or DQB1 antigen/allele mismatch

HLA-matching must be based on results of high resolution typing at HLA-A, -B, -C, -DRB1, and -DQ. If the patient is homozygous at the mismatch HLA class I locus or II locus, the donor must be heterozygous at that locus and one allele must match the patient (i.e., patient is homozygous A*01:01 and donor is heterozygous A*01:01, A*02:01)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-09-22 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary-Elizabeth Percival, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Chemotherapy, HCT): All patients enrolled received bridge chemotherapy prior to anticipated allogeneic hematopoietic cell transplantation (HCT). Patients received G-CLAM chemotherapy (consisting of G-CSF, mitoxantrone, cladribine, and cytarabine). HCT conditioning consisted of fludarabine and melphalan, with total body irradiation for patients over age 55 or with significant co-morbidities. HCT was to be received within 60 days of starting G-CLAM chemotherapy.
Period: Overall Study
Arm/Group | Treatment (Chemotherapy, HCT)
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Chemotherapy, HCT)
Number analyzed (Participants) | 30
Age, Customized [Median (Full Range); unit: years] | 56.5 [28 to 69]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 18
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 27
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 0
  White | 26
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30
High-Grade Myeloid Diagnosis [Count of Participants; unit: Participants]
  Acute myeloid leukemia (AML) | 29
  Myelodysplastic syndrome excess blasts 2 (MDS EB-2) | 1
Disease Status [Count of Participants; unit: Participants]
  Relapsed | 16
  Refractory | 14
Treatment Related Mortality Score [Median (Full Range); unit: units on a scale (0-100)] — Our institution defines TRM as death within 28 days from initiation of chemotherapy based on the observation that the risk of death declines once 4 weeks has elapsed from treatment start. A calculation is used to predict TRM using patient's age, performance status, if they have secondary AML, albumin, creatinine, platelet count, white blood cell count, and peripheral blood blast percentage. The higher the TRM score, the higher the risk of TRM. Calculator and table of relationship between TRM score and TRM probability found here: https://cstaging.fhcrc-research.org/TRM/Default.aspx
  units on a scale (0-100) | 2.33 [0.57 to 8.2]
ELN 2017 Risk Stratification [Count of Participants; unit: Participants]
  Favorable | 5
  Intermediate | 10
  Adverse | 15
Prior Lines of Therapy [Median (Full Range); unit: Number of prior treatment regimens] | 2 [1 to 3]
Duration of First Complete Remission [Median (Full Range); unit: Months] — The length of time, in months, between achieving a complete remission after initial chemotherapy and relapse.
  Months | 2 [0 to 31]

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Early Allogeneic Hematopoietic Cell Transplant Assessed by Enrollment and Incidence of Early Transplant
Description: Success will be defined as enrollment of at least 30 patients with transplants occurring in 15 of these 30 (50%) within 60 days of enrollment or start of induction chemotherapy with G-CLAM, whichever is earlier.
Time Frame: Up to 60 days after start of chemotherapy
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Chemotherapy, HCT)
Number analyzed (Participants) | 30
Participants
  Received allogeneic HCT on study within 60 days (feasibility success) | 9
  Did not receive allogeneic HCT on study within 60 days (feasibility failure) | 21

2. Primary Outcome: Feasibility of Early Allogeneic Hematopoietic Cell Transplant Assessed by Relapsed-free Survival 6 Months After Transplant
Description: Success will be defined as observing a 40% of higher 6-month relapse-free survival among patients who received early transplant on study.
Time Frame: 6 months after early allogeneic HCT on study
Population: Nine subjects received allogeneic HCT on study, however one subject died shortly after HCT and was not including in this analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Received Early Allogeneic HCT on Study: Patients who received an allogeneic hematopoietic peripheral blood stem cell transplantation within 60 days of bridge chemotherapy on study.
Arm/Group | Received Early Allogeneic HCT on Study
Number analyzed (Participants) | 9
Participants
  No relapse within 6 months post-HCT (feasibility success): number analyzed (Participants) | 8
  No relapse within 6 months post-HCT (feasibility success) | 6
  Relapse within 6 months post-HCT (feasibility failure): number analyzed (Participants) | 8
  Relapse within 6 months post-HCT (feasibility failure) | 2

3. Secondary Outcome: Response Assessments After Early Allogeneic Hematopoietic Cell Transplant, Day 28
Description: Complete Remission (CR), defined as <5% blasts in bone marrow with hematologic recovery (ANC>1000/ul and platelets >100,000/ml).
  CRi, defined as complete remission with insufficient hematologic recovery (ANC<1000/ul or platelets<100,000/ul).
  CRp, defined as complete remission but platelets <100,000/ul. Minimal residual disease (MRD), defined as any detectable disease by flow cytometry, cytogenetics, FISH or PCR in a patient otherwise fulfilling remission criteria.
  Morphologic leukemia-free state (MLFS), defined as <5% blasts in bone marrow with no hematologic recovery.
  Relapse, defined as >5% blasts in bone marrow, flow cytometry, or manual differential; OR treatment for active relapsed disease.
Time Frame: Approximately 28 days after early allogeneic HCT
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- Received Allogeneic HCT on Study: Patients who received an allogeneic hematopoietic peripheral blood stem cell transplantation within 60 days of bridge chemotherapy on study.
Arm/Group | Received Allogeneic HCT on Study
Number analyzed (Participants) | 9
Participants
  CR with MRD: number analyzed (Participants) | 8
  CR with MRD | 0
  CR without MRD: number analyzed (Participants) | 8
  CR without MRD | 7
  CRi with MRD: number analyzed (Participants) | 8
  CRi with MRD | 0
  CRi without MRD: number analyzed (Participants) | 8
  CRi without MRD | 1
  MLFS with MRD: number analyzed (Participants) | 8
  MLFS with MRD | 0
  MLFS without MRD: number analyzed (Participants) | 8
  MLFS without MRD | 0
  Relapse: number analyzed (Participants) | 8
  Relapse | 0

4. Secondary Outcome: Response Assessments After Early Allogeneic Hematopoietic Cell Transplant, Day 84
Description: as for outcome 3
Time Frame: Approximately 84 days after early allogeneic HCT
Population: Nine subjects received allogeneic HCT on study, however one subject died shortly after HCT and was not included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Received Allogeneic HCT on Study
Number analyzed (Participants) | 9
Participants
  CR with MRD: number analyzed (Participants) | 8
  CR with MRD | 0
  CR without MRD: number analyzed (Participants) | 8
  CR without MRD | 4
  CRi with MRD: number analyzed (Participants) | 8
  CRi with MRD | 0
  CRi without MRD: number analyzed (Participants) | 8
  CRi without MRD | 2
  MLFS with MRD: number analyzed (Participants) | 8
  MLFS with MRD | 0
  MLFS without MRD: number analyzed (Participants) | 8
  MLFS without MRD | 0
  Relapse: number analyzed (Participants) | 8
  Relapse | 2

5. Secondary Outcome: Relapse-free Survival (RFS) Among Patients Who Received Early Transplant
Description: Relapse-free survival among patients who received early allogeneic HCT on study as estimated with the Kaplan-Meier method.
Time Frame: Up to 100 days post-transplant
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Received Allogeneic HCT on Study
Number analyzed (Participants) | 9
Percentage of participants | 91 [85 to 100]

6. Secondary Outcome: Relapse-free Survival (RFS) Among Patients Who Received Early Transplant
Description: as for outcome 5
Time Frame: Up to 6 months post-transplant
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Received Allogeneic HCT on Study
Number analyzed (Participants) | 9
Percentage of participants | 82 [62 to 100]

7. Secondary Outcome: Event-free Survival (EFS) Among Patients Who Received Early Transplant
Description: Event-free survival among patients who received early allogeneic HCT on study as estimated with the Kaplan-Meier method. Events included death, relapse, and grade 3-4 acute graft vs host disease.
Time Frame: Up to 100 days post-transplant
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Received Allogeneic HCT on Study
Number analyzed (Participants) | 9
Percentage of participants | 91 [85 to 100]

8. Secondary Outcome: Event-free Survival (EFS) Among Patients Who Received Early Transplant
Description: as for outcome 7
Time Frame: Up to 6 months post-transplant
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Received Allogeneic HCT on Study
Number analyzed (Participants) | 9
Percentage of participants | 82 [62 to 100]

9. Secondary Outcome: Overall Survival (OS) Among Patients Who Received Early Transplant.
Description: Overall survival among patients who received early allogeneic HCT on study as estimated with the Kaplan-Meier method.
Time Frame: Up to 100 days post-transplant
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Received Allogeneic HCT on Study
Number analyzed (Participants) | 9
Percentage of participants | 91 [85 to 100]

10. Secondary Outcome: Overall Survival (OS) Among Patients Who Received Early Transplant.
Description: Overall survival among patients who received early allogeneic HCT on study as estimated with the Kaplan-Meier method.
Time Frame: Up to 6 months post-transplant
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Received Allogeneic HCT on Study
Number analyzed (Participants) | 9
Percentage of participants | 82 [62 to 100]

11. Secondary Outcome: Overall Survival (OS) Among Patients Who Did Not Receive Early Transplant
Description: Overall survival among patients who did not receive early allogeneic HCT on study as estimated with the Kaplan-Meier method.
Time Frame: Up to 100 days after induction day 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Did Not Receive Allogeneic HCT on Study: Patients who did not receive an allogeneic hematopoietic peripheral blood stem cell transplantation within 60 days of bridge chemotherapy on study.
Arm/Group | Did Not Receive Allogeneic HCT on Study
Number analyzed (Participants) | 21
Percentage of participants | 75 [60 to 97]

12. Secondary Outcome: Overall Survival (OS) Among Patients Who Did Not Receive Early Transplant
Description: as for outcome 11
Time Frame: Up to 6 months after induction day 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Did Not Receive Allogeneic HCT on Study
Number analyzed (Participants) | 21
Percentage of participants | 62 [44 to 87]

13. Secondary Outcome: Acute Graft Versus Host Disease Among Patients Who Received Early Transplant
Description: Acute graft versus host disease (graded II, III, or IV) among patients who received early allogeneic HCT on study.
Time Frame: At day 100
Measure: Count of Participants; unit: Participants
Arm/Group | Received Allogeneic HCT on Study
Number analyzed (Participants) | 9
Participants | 0

14. Secondary Outcome: Treatment Related Mortality Among Patients Who Received Early Transplant vs Patients Who Did Not Receive Early Transplant
Description: Treatment related mortality calculated among patients who received early allogeneic HCT on study vs patients who did not receive early transplant on study.
Time Frame: At day 100
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Received Allogeneic HCT on Study | Did Not Receive Allogeneic HCT on Study
Number analyzed (Participants) | 9 | 21
Percentage of participants | 9 [0 to 27] | 23.8 [5 to 43]
Statistical Analysis 1: Comparison: Received Allogeneic HCT on Study vs Did Not Receive Allogeneic HCT on Study; Test type: Other; p = 0.18, Wilcoxon (Mann-Whitney)

15. Secondary Outcome: Factors That Distinguish Patients Who Received Early Transplant From Those Who Did Not - TREATMENT RELATED MORTALITY
Description: Patients who receive early transplant will be compared to those that don't using the Wilcoxon rank sum test for the quantitative variable of treatment-related mortality (TRM). This outcome measure is intended to report a predicted TRM score assessed at the time of feasibility evaluation. The TRM score is used to measure "treatment-related mortality," or likelihood of death within 28 days of initiation of induction chemotherapy for patients with AML. The score is normalized from 0 to 100, so that a score of 0 demonstrates the patient has a very low likelihood of TRM and a score of 100 a very high likelihood of death. A calculation is used to predict TRM using age, performance status, if they have secondary AML, albumin, creatinine, platelet count, white blood cell count, and peripheral blood blast percentage. The higher the TRM score, the higher the risk of TRM. Calculator and table of relationship between TRM score and TRM probability found here: https://trmcalculator.fredhutch.org/.
Time Frame: From time of subject's study enrollment to time of subject's feasibility success assessment (i.e. when subject received transplant within 60 days or when it was determined subject would not proceed with transplant on study)
Population: Only 18 of the 21 patients who did not receive an allogeneic hematopoietic peripheral blood stem cell within 60 days of bridge chemotherapy on study were analyzed.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Received Allogeneic HCT on Study | Did Not Receive Allogeneic HCT on Study
Number analyzed (Participants) | 9 | 18
units on a scale | 2.15 [0.61 to 3.67] | 3.045 [0.57 to 8.2]
Statistical Analysis 1: Comparison: Received Allogeneic HCT on Study vs Did Not Receive Allogeneic HCT on Study; Test type: Other; p = 0.18, Wilcoxon (Mann-Whitney)

16. Secondary Outcome: Factors That Distinguish Patients Who Received Early Transplant From Those Who Did Not - GENDER
Description: Patients who receive early transplant will be compared to those that don't using the Fisher's exact test for the categorical variables of gender.
Time Frame: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Received Allogeneic HCT on Study | Did Not Receive Allogeneic HCT on Study
Number analyzed (Participants) | 9 | 21
Participants
  Female | 8 | 10
  Male | 1 | 11
Statistical Analysis 1: Comparison: Received Allogeneic HCT on Study vs Did Not Receive Allogeneic HCT on Study; Test type: Other; p = 0.049, Fisher Exact

17. Secondary Outcome: Factors That Distinguish Patients Who Received Early Transplant From Those Who Did Not - AGE
Description: Patients who receive early transplant will be compared to those that don't using the Wilcoxon rank sum test for the quantitative variable of age.
Time Frame: as for outcome 15
Measure: Median (Full Range); unit: years
Arm/Group | Received Allogeneic HCT on Study | Did Not Receive Allogeneic HCT on Study
Number analyzed (Participants) | 9 | 21
years | 55 [36 to 67] | 57 [28 to 69]
Statistical Analysis 1: Comparison: Received Allogeneic HCT on Study vs Did Not Receive Allogeneic HCT on Study; Test type: Other; p = 0.77, Wilcoxon (Mann-Whitney)

18. Secondary Outcome: Demonstrate the Feasibility of Collecting Patient-reported Outcomes for Trial Participants
Description: The amount of returned patient-reported outcome questionnaires will be summarized for each collection timepoint using percent collection from surviving patients for PRO timepoints.
Time Frame: Up to 12 months post-HCT
Population: The number analyzed in each of the rows below represent the patients alive at that timepoint who were due to complete a survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Chemotherapy, HCT)
Number analyzed (Participants) | 30
Participants
  Enrollment PROs returned | 27
  Post G-CLAM PROs returned | 23
  Pre-HCT PROs returned: number analyzed (Participants) | 9
  Pre-HCT PROs returned | 8
  6 months post-HCT PROs returned: number analyzed (Participants) | 7
  6 months post-HCT PROs returned | 4
  12 months post-HCT PROs returned: number analyzed (Participants) | 5
  12 months post-HCT PROs returned | 3

19. Secondary Outcome: Demonstrate the Feasibility of Collecting Resource Utilization Data for Trial Participants
Description: The amount of days of hospitalization (the major driver of costs within the first year) will be collected for resource utilization.
Time Frame: Within the first year of induction chemotherapy on study
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Treatment (Chemotherapy, HCT)
Number analyzed (Participants) | 30
days | 49 [32 to 56]

ADVERSE EVENTS:
Time Frame: Serious adverse events monitoring started Day 1 of G-CLAM therapy or the date of consent, whichever date came first, until: • Up to day 100 after transplant, for subjects who are "successes" • The date the subject is off-study, for subjects who are "failures" and did not receive transplant within 60 days All-cause mortality monitoring started on Day 1 of G-CLAM therapy or the date of consent, whichever date came first, to 6-months post transplant.
Description: Other (not including serious) adverse events were not collected and reported.
Groups:
- Post-Chemotherapy: All patients enrolled received bridge chemotherapy prior to anticipated allogeneic hematopoietic cell transplantation (HCT). Patients received G-CLAM chemotherapy (consisting of G-CSF, mitoxantrone, cladribine, and cytarabine).
- Post-Transplant: Allogeneic peripheral blood stem cell transplant with reduced-intensity conditioning regimen consisted of fludarabine and melphalan, with total body irradiation for subjects over age 55. Prophylaxis for acute graft-vs-host-disease was mycophenylate mofetil (MMF), cyclosporine, and sirolimus.
Arm/Group | Post-Chemotherapy | Post-Transplant
All-Cause Mortality (participants affected / at risk) | 5/30 | 2/9
Serious Adverse Events (participants affected / at risk) | 30/30 | 9/9
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Post-Chemotherapy (N=30) | Post-Transplant (N=9)
Headache (Nervous system disorders) | 3 (3) | 0 (0)
Intracranial lesions (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 0 (0)
Stroke (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 2 (2)
Hallucinations (Psychiatric disorders) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 2 (2)
Hypotension (Vascular disorders) | 2 (3) | 1 (1)
Typhlitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bowel perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Nausea with vomiting (Gastrointestinal disorders) | 0 (0) | 3 (4)
Mucositis (Gastrointestinal disorders) | 0 (0) | 6 (6)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Alanine aminotransferase increased (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Alkaline phosphatase increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Blood bilirubin increased (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (2)
Acute hypoxemic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (2)
Diffuse aveolar hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Heart failure (Cardiac disorders) | 2 (2) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Allergic reaction (Immune system disorders) | 2 (2) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 1 (1)
Lung infection (Infections and infestations) | 6 (7) | 0 (0)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2)
Skin infection (Infections and infestations) | 3 (3) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 14 (17) | 8 (8) — No source identified.
Bacteremia (Infections and infestations) | 12 (16) | 2 (2)
Sepsis (Infections and infestations) | 2 (3) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Liver fibrosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Ejection fraction decreased (Investigations) | 1 (1) | 0 (0)
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 (0) | 2 (2)
Edema in limbs (General disorders) | 0 (0) | 1 (1)
Multi-organ failure (General disorders) | 1 (1) | 0 (0)
Deconditioning/poor functional status (General disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Some patients did not move on with transplant on study within 60 days of chemotherapy due to issues with scheduling pre-transplant evaluations, donor searches, and donor availability which caused delays. Some patients were also taken off this study to enroll onto other, more appropriate transplant clinical trials.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-25): https://cdn.clinicaltrials.gov/large-docs/72/NCT02756572/Prot_SAP_001.pdf